CLINICAL TRIAL: NCT06090773
Title: Characteristics of Renal Blood Flow in AKI Patients With Sepsis and Its Clinical Significance
Brief Title: Characteristics of Renal Blood Flow in AKI Patients in ICU and Its Clinical Significance
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-PUMCH-A-218
Record Dates: First submitted 2023-10-14; First posted 2023-10-19 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Acute Kidney Injury; Renal Artery Blood Flow; Renal Venous Return; Renal Microcirculation
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acute kidney injury: Patients with acute injuries in ICU patients.
- Patients with non-acute kidney injury: ICU patients without acute injury patients.

SUMMARY:
To study the changes in the renal artery and renal vein with renal cortical and medullary microcirculatory blood flow in patients with sepsis; to study the relationship between renal arteriolar and renal vein with renal cortical and medullary microcirculatory blood flow and renal function; and to find the value of ultrasonographic assessment of renal blood flow indices for evaluating prognosis in patients with sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-85 years old; Control group: patients with non-acute kidney injury after ICU general surgery; Observation group: patients who met the diagnostic criteria of AKI: Scr elevation ≥26.5 umol/L within 48h; Scr elevation exceeding 1.5 times and more than the basal value within 7d; and decrease in urine output (<0.5 ml/kg/h) with a duration of 6h or more.

Exclusion Criteria:

* Those who did not meet the inclusion criteria or refused to be enrolled; patients with underlying end-stage renal disease or requiring long-term dialysis; renal transplant patients; patients with other underlying systemic diseases causing renal dysfunction (SCr > 88.4 umol/L); those who were unable to obtain a clear renal ultrasound view; those with suspected contrast allergy; those with pulmonary arterial systolic blood pressure ≥ 90 mm Hg; and those who were pregnant or breastfeeding women.

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Age between 18-85 years old; Control group: patients with non-acute kidney injury after ICU general surgery; Observation group: patients who met the diagnostic criteria of AKI: Scr elevation ≥26.5 umol/L within 48h; Scr elevation exceeding 1.5 times and more than the basal value within 7d; and decrease in urine output (<0.5 ml/kg/h) with a duration of 6h or more.
Sampling Method: Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
30-day major renal adverse events | 30-day
  Follow-up of patients with prognostic indicators of renal function within 30 days of enrolment, such as blood creatinine and the need for renal replacement therapy.
Renal artery blood flow | Day 1,Day 3,Day 5, Day 7
  Ultrasound assessment of renal artery resistance index, and renal artery blood flow.
Renal venous return | Day 1,Day 3,Day 5, Day 7
  Ultrasonographic assessment of renal venous reflux profiles.
renal microcirculation | Day 1,Day 3,Day 5, Day 7
  Evaluation of renal microcirculation by ultrasonography.

CONTACTS AND LOCATIONS:
Locations (1):
- Rongping Chen, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No